CLINICAL TRIAL: NCT05426967
Title: ADEPT: Adaptive Trial for the Treatment of Depressive Symptoms Associated With Concussion Using Repetitive Transcranial Magnetic Stimulation Protocols
Brief Title: rTMS for Military TBI-related Depression
Acronym: ADEPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USUHS-2020-050
Record Dates: First submitted 2022-03-07; First posted 2022-06-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Depressive Symptoms; Mild Traumatic Brain Injury; Concussion
Keywords: Transcranial Magnetic Stimulation (TMS); Depressive Symptoms; Concussion; Mild Traumatic Brain Injury (TBI); Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Depression; Brain Concussion | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Bayesian-adaptive trial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm 1 (Experimental): Active rTMS/Individualized Connectome Targeting (ICT)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Arm 2 (Experimental): Active rTMS/resting state functional MRI (rsfMRI)-based targeting
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Arm 3 (Sham Comparator): Sham rTMS
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Active rTMS
  Arms: Arm 1; Arm 2
Device: Sham rTMS — Sham comparator to active rTMS
  Arms: Arm 3

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, and tolerability of two dorsolateral prefrontal cortex (DLPFC) repetitive transcranial magnetic stimulation (rTMS) protocols to alleviate symptoms of depression in United States (U.S.) military service members and veterans with a history of concussion/mild traumatic brain injury (TBI).

DETAILED DESCRIPTION:
In United States Military personnel, rates of depression may increase after mild traumatic brain injury, or concussion. rTMS may hold a therapeutic potential for alleviating symptoms of depression after concussion. This study is a randomized, double-blind, Bayesian adaptive trial aimed at determining the safety, efficacy, and tolerability of individualized connectome targeted (ICT)-accelerated intermittent Theta Burst Stimulation (aiTBS) and scalp-targeted aiTBS for the treatment of depressive symptoms in a properly powered sample of current and former US military service members with a history of concussion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 at the time of consent. Older individuals will not be enrolled in this initial trial for reasons of safety and expected reduced efficacy.
* Current or former US military service member eligible for care at a Military Treatment Facility (MTF) or Veterans Administration Medical Center (VAMC.)
* Able to provide written, informed consent in English .
* Self-reported or medically diagnosed history of concussion (synonymous with "mild TBI.") >6 months, but <26 years prior to consent, defined based on the DoD/VA definition:

  1. Positive Loss of Consciousness of <30 minutes as confirmed by the TBI Screener and/or medical records and/or;
  2. Positive Alteration of Consciousness of <24 hours as confirmed by the TBI Screener and/or medical records and/or;
  3. Positive Post-traumatic Amnesia of 0 to 1 day as confirmed by the TBI Screener and/or medical records.

     * Note: Neuroimaging data or documentation from medical records is not required.
* Baseline MADRS >13 at the time of screening indicating at least mild-moderate depressive symptoms.
* Maintained a steady psychotropic medication regimen for six weeks and a steady behavioral therapy regimen for twelve weeks prior to enrollment in the study.
* Female participants with child-bearing potential must agree to use an effective method of birth control during the course of the study.
* Under the care of a primary care and/or behavioral health provider.

Exclusion Criteria:

* Elevated risk of seizures at the time of rTMS including any of the following:

  1. History of unprovoked seizures.
  2. History of seizure within 24 hours of sustaining a concussion(s) or other head injury regardless of whether it was determined to have been related to concussion.
  3. Family history of two or more unprovoked seizures in a first degree relative (parent, sibling, or child).
  4. History of Moderate, Severe, or Penetrating TBI based on TBI Screener and/or medical records.
  5. Intracranial lesion (such as intracranial tumor or intraparenchymal hemorrhage) that, in the opinion of the investigators, would increase seizure risk.
  6. Currently taking medication or other substances (such as tricyclic antidepressants or neuroleptics) that, in the opinion of the investigator, lowers the seizure threshold.
* Contraindications to awake 3T MRI without contrast at the time of the Baseline MRI according to site radiology department criteria.
* Severe claustrophobia interfering with medication/sedation-free 3T closed-bore MRI.
* Intracranial lesion that would produce an artifact that would compromise the integrity of rsfMRI data.
* History of severe or recent uncontrolled heart disease.
* Presence of a cardiac pacemaker or intracardiac lines.
* Any implant, prosthesis or other permanent alteration of the body (such as implanted neurostimulators and medication pumps) that, in the opinion of the investigator, would be unsafe with MRI or TMS or that would produce an artifact that would compromise the integrity of data.
* Presence of rapidly progressive illnesses such as late-stage cancer, neurodegenerative conditions, major organ failure, etc.
* History of Bipolar Disorder or Schizophrenia Spectrum Disorders.
* Current evidence of substance-induced mood disorder, active psychosis, or depression secondary to general medical illness other than TBI.
* Severe or uncontrolled substance use.
* Concomitant or lifetime history of receiving open-label TMS, due to issues preserving blinding.
* Concomitant or recent history (within 12 weeks prior to enrollment) of receiving other neurostimulatory treatment, including but not limited to transcranial direct current (tDCS), transcranial alternating current (tACS), alpha stim, or electroconvulsive therapy.
* Suicide attempt within six months prior to enrollment.
* Right upper extremity amputation or other condition precluding left motor threshold calibration.
* Unable to complete timeline of study (e.g., planned hospitalization partway through the study period.)
* Prisoner, or other legally restricted freedom of movement and participation.
* Any other considerations that, in the opinion of the investigators, may adversely affect participant safety, participation, or the scientific validity of the data being collected (e.g., erratic or unreliable responses, inconsistent communication, inability to remain on a steady neurotropic medication and/or behavioral therapy regimen over the course of the Randomization phase of the study.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Scores | Baseline to post-intervention, within 10 working days of the final rTMS session
  Change in Montgomery-Asberg Depression Rating Scale scores from baseline to post-intervention between groups. The Scale is designed to measure depression severity and consists of 10 items, each of which is scored on a Likert scale from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Scores in a Subgroup | Baseline to post-intervention, within 10 working days of the final rTMS session
  Change in Montgomery-Asberg Depression Rating Scale scores between groups from Baseline to post-intervention in participants who complete ≥80% of rTMS sessions. The Scale is designed to measure depression severity and consists of 10 items, each of which is scored on a Likert scale from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) Scores from Baseline to 6-month follow-up | Baseline to 6 months
  Change in Montgomery-Asberg Depression Rating Scale scores from baseline to 6-month follow-up between groups. The Scale is designed to measure depression severity and consists of 10 items, each of which is scored on a Likert scale from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Comparison of Treatment Response or Remission in Montgomery-Asberg Depression Rating Scale (MADRS) Scores | Baseline to post-intervention, within 10 working days of the final rTMS session
  Comparison of proportion of participants in each condition achieving treatment response ≥50% improvement in MADRS) or remission (MADRS ≤10)
Comparison of Duration of Remission of Depressive Symptoms in Montgomery-Asberg Depression Rating Scale (MADRS) Scores | Follow-up Period, from 1-6 months after the final rTMS session
  Comparison of duration of remission of depressive symptoms in Montgomery-Asberg Depression Rating Scale (MADRS) Scores between groups assessed monthly during follow-up
Comparison of Frequency of Adverse Events | Baseline to post-intervention, within 10 working days of the final rTMS session
  Comparison of AEs between groups

SECONDARY OUTCOMES:
Comparison of Change in Inventory of Depressive Symptomatology-Self Report (IDS-SR) Scores from Baseline to post-intervention | Baseline to post-intervention, within 10 working days of the final rTMS session
  Change in Inventory of Depressive Symptomatology-Self Report scores between groups. The Report is a 30-item self-report depressive symptom severity rating scale, with each question on a scale of 0 to 4; and a score range between 0 to 84, with a higher score reflecting higher symptom severity in depression.
Comparison of Change in Symptoms of Major Depressive Disorder Scale (SMDDS) Scores from Baseline to Post-intervention | Baseline to post-intervention, within 10 working days of the final rTMS session
  Change in Symptoms of Major Depressive Disorder Scale scores between groups. The Scale is a 16-question scale, with each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always"); the total score ranges from 0 to 60 with a higher score indicating more severe depressive symptomatology.
Comparison of Change in Inventory of Depressive Symptomatology-Self Report (IDS-SR) Scores from Baseline to 6-month follow-up | Baseline to 6-month follow-up
  Change in Inventory of Depressive Symptomatology-Self Report scores between groups. The Report is a 30-item self-report depressive symptom severity rating scale, with each question on a scale of 0 to 4; and a score range between 0 to 84, with a higher score reflecting higher symptom severity in depression
Comparison of Change in Symptoms of Major Depressive Disorder Scale (SMDDS) Scores from Baseline to 6-month follow-up | Baseline to 6-month follow-up
  Change in Symptoms of Major Depressive Disorder Scale scores between groups. The Scale is a 16-question scale, with each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always"); the total score ranges from 0 to 60 with a higher score indicating more severe depressive symptomatology.
Comparison of Change in TBI Quality of Life Scale (TBI-QOL) Subtest Scores from Baseline to Post-intervention | Baseline to post-intervention, within 10 working days of the final rTMS session
  Change in subtest scores between groups Anxiety ranges Raw Score (RS) 10-50, T-score 36.0-85.1; higher = worse Communication ranges RS 9-45, T-score 12.8-67.2; higher = better Depression ranges RS 10-50, T-score 38.3-82.6; higher = worse Emotional & Behavioral Dyscontrol ranges RS 10-50, T-score 33.1-84.6; higher = worse Executive Function range RS 10-50, T-score 12.3-58.0; higher = better Fatigue ranges RS 10-50, T-score 32.7-80.7; higher = worse General Concerns ranges RS 10-50, T-score 17.3-59.6; higher = better Grief - Loss ranges RS 9-45, T-score 32.9-75.0; higher = worse Headache ranges RS 10-50, T-score 38.9-72.6; higher = worse Independence ranges RS 8-40, T-score 21.2-66.2; higher = better Pain Interference ranges RS 10-50, T-score 40.4-78.8; higher = worse Resilience ranges RS 10-50, T-score 15.3-69.2; higher = better Self-Esteem ranges RS 10-50, T-score 20.0-64.9; higher = better Cognitive Function ranges RS 8-40, T-score 22.5-67.0; higher = better
Comparison of Change in TBI Quality of Life Scale (TBI-QOL) Subtest Scores from Baseline to 6-month follow-up | Baseline to 6-month follow-up
  Change in subtest scores between groups Anxiety ranges Raw Score (RS) 10-50, T-score 36.0-85.1; higher = worse Communication ranges RS 9-45, T-score 12.8-67.2; higher = better Depression ranges RS 10-50, T-score 38.3-82.6; higher = worse Emotional & Behavioral Dyscontrol ranges RS 10-50, T-score 33.1-84.6; higher = worse Executive Function range RS 10-50, T-score 12.3-58.0; higher = better Fatigue ranges RS 10-50, T-score 32.7-80.7; higher = worse General Concerns ranges RS 10-50, T-score 17.3-59.6; higher = better Grief - Loss ranges RS 9-45, T-score 32.9-75.0; higher = worse Headache ranges RS 10-50, T-score 38.9-72.6; higher = worse Independence ranges RS 8-40, T-score 21.2-66.2; higher = better Pain Interference ranges RS 10-50, T-score 40.4-78.8; higher = worse Resilience ranges RS 10-50, T-score 15.3-69.2; higher = better Self-Esteem ranges RS 10-50, T-score 20.0-64.9; higher = better Cognitive Function ranges RS 8-40, T-score 22.5-67.0; higher = better
Comparison of Change in PTSD Checklist for DSM-5 (PCL-5) Scores from Baseline to Post-intervention | Baseline to post-intervention, within 10 working days of the final rTMS session
  Change in PTSD Checklist for DSM-5 scores between groups. The Checklist is a self-reported measure of PTSD symptom severity, with a score range of 0-84 in which a higher score represents greater severity.
Comparison of Change in PTSD Checklist for DSM-5 (PCL-5) Scores from Baseline to 6-month Follow-up | Baseline to 6-month follow-up
  Change in PTSD Checklist for DSM-5 scores between groups. The Checklist is a self-reported measure of PTSD symptom severity, with a score range of 0-84 in which a higher score represents greater severity.
Compliance Assessment | Post-intervention, within 10 working days of the final rTMS session
  Proportion of participants who achieve at least 80% compliance, defined as having completed ≥16 rTMS sessions
Comparison of Change in rsfMRI Connectivity from Baseline to Post-intervention | Baseline to post-intervention, within 10 working days of the final rTMS session
  Compare change in rsfMRI connectivity, focusing on brain networks relevant to mood regulation between groups
Comparison of Change in rsfMRI Connectivity from Baseline to 6-month Follow-up | Baseline to 6-month follow-up
  Compare change in rsfMRI connectivity, focusing on brain networks relevant to mood regulation between groups

CONTACTS AND LOCATIONS:
Overall Officials: David L Brody, MD, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, California
  - William Beaumont Army Medical Center, Fort Bliss, Texas
  - Alexander T. Augusta Military Medical Center, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Identifier-free data sets may also be shared with the Federal Interagency Traumatic Brain Injury Research (FITBIR) Data Repository
Time Frame: After study completion, data sets will be de-identified and shared with the repositories. De-identified data sets will be stored in the repositories indefinitely.
Access Criteria: Access to FITBIR will follow FITBIR Access Criteria.
URL: http://fitbir.nih.gov/content/access-data

REFERENCES:
- [Derived] Oberman LM, Penafiel AI, Dieterich R, Phan CT, Chou YY, Pham DL, Adamson MM, Hines CE, Rezaee Z, Deng ZD, Pal H, Lisanby SH, Brody DL. Adaptive trial for the treatment of depressive symptoms associated with concussion using accelerated intermittent theta burst stimulation (ADEPT): rationale, design and methods. Front Neurol. 2025 Jun 13;16:1605157. doi: 10.3389/fneur.2025.1605157. eCollection 2025. PMID 40584527